CLINICAL TRIAL: NCT05431712
Title: Impact of Donor-Specific Antibodies in (Highly-) Immunized Living Donor Kidney Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Annelies de Weerd, MD, PhD, MD, PhD, Principal investigator, Erasmus Medical Center
Other Study IDs: MEC-2021-0357
Record Dates: First submitted 2022-06-14; First posted 2022-06-24 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- DSA+: Patients with pre-transplantation detected donor-specific antibodies, with Luminex Single Antigen Bead analysis.
- PRA+: Immunized controls without DSAs pre-transplantation, with equal peak PRA levels and donor/recipient age as the DSA+ group.
- PRA-: Non-immunized controls without DSAs pre-transplantation, with a peak PRA of less than 6%, with equal donor/recipient age as the DSA+ group.

SUMMARY:
Kidney transplantation is the preferred treatment for end-stage renal disease. Alongside limited availability of donors, rejection and premature graft loss are main barriers to kidney transplantation. Donor-specific antibodies pre-transplantation may arise due to to prior solid organ transplantation, pregnancy or blood transfusions. Their presence is considered a risk of graft failure. The impact of DSA is differently reported in literature, also according to the technique by which DSA have been measured. Techniques such as the complement-dependent cytotoxicity crossmatch, the immunofluorescence crossmatch and the Luminex Single Antigen Bead have different sensitivities for detecting DSA.

Historically, our kidney transplant program has been advocating living donor transplantation and as a result the majority of transplantations are with a living donor. In this context and in the absence of a compatible living donor, pretransplant DSA have not been considered an absolute contra-indication for transplantation. The aim of the current study is to determine the effect of DSAs on rejection and death-censored graft survival in living donor kidney transplantation.

Participants are adults who underwent a living donor kidney transplantation between 2010 and 2019 in the presence of DSA. Control subjects are both immunized and non-immunized kidney transplant recipients in the same period.

This is a retrospective, case control study. Death-censored graft survival is analyzed for all patients and compared by presence of DSA and other predicting variables, such as immunization level, age, sex and HLA mismatches. Furthermore, biopsy proven rejection, patient survival, kidney function, length of hospital stay and proteinuria are analyzed.

Also, a predefined subgroup analysis is performed in the DSA positive patients. These are compared according to amount, strength and HLA-class of DSAs.

ELIGIBILITY:
Inclusion Criteria:

* Pre-transplantation donor-specific antibodies in Luminex Single Antigen Bead analysis.
* Age 18 years or older

Exclusion Criteria:

* Desensitization treatment for a current or historic positive CDC-crossamtch

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive kidney transplant recipients in the period 2010-2019, who had pre-transplantation donor-specific antibodies detected in Luminex Single Antigen Bead analysis.
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Death-censored graft survival | 4-12 years
  Amount of patients who were alive with a functioning graft, divided by all alive included patients at different moments in time.

SECONDARY OUTCOMES:
Patient survival | 4-12 years
  Amount of patients alive, divided by total amount of included patients at different moments in time.
Biopsy proven rejection | 4-12 years
  Amount of patients with a pathologically confirmed rejection.
Hospital admission days | first year post-transplantation
  Number of days that the patient spent admitted to the hospital.
Renal function | first year post-transplantation
  Estimated Glomerular Filtration Rate (eGFR)
Proteinuria | first year post-transplantation
  Grams of protein per 1 liter of urine.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chung BH, Choi BS, Oh EJ, Park CW, Kim JI, Moon IS, Kim YS, Yang CW. Clinical impact of the baseline donor-specific anti-human leukocyte antigen antibody measured by Luminex single antigen assay in living donor kidney transplant recipients after desensitization therapy. Transpl Int. 2014 Jan;27(1):49-59. doi: 10.1111/tri.12199. Epub 2013 Oct 25. PMID 24118413
- [Background] Betjes MGH, Sablik KS, Otten HG, Roelen DL, Claas FH, de Weerd A. Pretransplant Donor-Specific Anti-HLA Antibodies and the Risk for Rejection-Related Graft Failure of Kidney Allografts. J Transplant. 2020 Jan 29;2020:5694670. doi: 10.1155/2020/5694670. eCollection 2020. PMID 32099669
- [Background] Kamburova EG, Wisse BW, Joosten I, Allebes WA, van der Meer A, Hilbrands LB, Baas MC, Spierings E, Hack CE, van Reekum FE, van Zuilen AD, Verhaar MC, Bots ML, Drop ACAD, Plaisier L, Seelen MAJ, Sanders JSF, Hepkema BG, Lambeck AJA, Bungener LB, Roozendaal C, Tilanus MGJ, Voorter CE, Wieten L, van Duijnhoven EM, Gelens M, Christiaans MHL, van Ittersum FJ, Nurmohamed SA, Lardy NM, Swelsen W, van der Pant KA, van der Weerd NC, Ten Berge IJM, Bemelman FJ, Hoitsma A, van der Boog PJM, de Fijter JW, Betjes MGH, Heidt S, Roelen DL, Claas FH, Otten HG. Differential effects of donor-specific HLA antibodies in living versus deceased donor transplant. Am J Transplant. 2018 Sep;18(9):2274-2284. doi: 10.1111/ajt.14709. Epub 2018 Apr 16. PMID 29464832
- [Background] Ziemann M, Altermann W, Angert K, Arns W, Bachmann A, Bakchoul T, Banas B, von Borstel A, Budde K, Ditt V, Einecke G, Eisenberger U, Feldkamp T, Gorg S, Guthoff M, Habicht A, Hallensleben M, Heinemann FM, Hessler N, Hugo C, Kaufmann M, Kauke T, Koch M, Konig IR, Kurschat C, Lehmann C, Marget M, Muhlfeld A, Nitschke M, Pego da Silva L, Quick C, Rahmel A, Rath T, Reinke P, Renders L, Sommer F, Spriewald B, Staeck O, Stippel D, Susal C, Thiele B, Zecher D, Lachmann N. Preformed Donor-Specific HLA Antibodies in Living and Deceased Donor Transplantation: A Multicenter Study. Clin J Am Soc Nephrol. 2019 Jul 5;14(7):1056-1066. doi: 10.2215/CJN.13401118. Epub 2019 Jun 18. PMID 31213508
- [Background] Orandi BJ, Garonzik-Wang JM, Massie AB, Zachary AA, Montgomery JR, Van Arendonk KJ, Stegall MD, Jordan SC, Oberholzer J, Dunn TB, Ratner LE, Kapur S, Pelletier RP, Roberts JP, Melcher ML, Singh P, Sudan DL, Posner MP, El-Amm JM, Shapiro R, Cooper M, Lipkowitz GS, Rees MA, Marsh CL, Sankari BR, Gerber DA, Nelson PW, Wellen J, Bozorgzadeh A, Gaber AO, Montgomery RA, Segev DL. Quantifying the risk of incompatible kidney transplantation: a multicenter study. Am J Transplant. 2014 Jul;14(7):1573-80. doi: 10.1111/ajt.12786. Epub 2014 Jun 9. PMID 24913913
- [Background] Orandi BJ, Luo X, Massie AB, Garonzik-Wang JM, Lonze BE, Ahmed R, Van Arendonk KJ, Stegall MD, Jordan SC, Oberholzer J, Dunn TB, Ratner LE, Kapur S, Pelletier RP, Roberts JP, Melcher ML, Singh P, Sudan DL, Posner MP, El-Amm JM, Shapiro R, Cooper M, Lipkowitz GS, Rees MA, Marsh CL, Sankari BR, Gerber DA, Nelson PW, Wellen J, Bozorgzadeh A, Gaber AO, Montgomery RA, Segev DL. Survival Benefit with Kidney Transplants from HLA-Incompatible Live Donors. N Engl J Med. 2016 Mar 10;374(10):940-50. doi: 10.1056/NEJMoa1508380. PMID 26962729
- [Background] Jordan SC, Lorant T, Choi J, Kjellman C, Winstedt L, Bengtsson M, Zhang X, Eich T, Toyoda M, Eriksson BM, Ge S, Peng A, Jarnum S, Wood KJ, Lundgren T, Wennberg L, Backman L, Larsson E, Villicana R, Kahwaji J, Louie S, Kang A, Haas M, Nast C, Vo A, Tufveson G. IgG Endopeptidase in Highly Sensitized Patients Undergoing Transplantation. N Engl J Med. 2017 Aug 3;377(5):442-453. doi: 10.1056/NEJMoa1612567. PMID 28767349